CLINICAL TRIAL: NCT04855916
Title: ABLE Exoskeleton vs KAFO Orthosis: Comparative Study of Gait Kinematics and Energy Efficiency in Patients With Spinal Cord Injury
Brief Title: KAFO Orthoses Versus the ABLE Exoskeleton
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ABLE Human Motion S.L. (Industry)
Collaborators: Hospital Asepeyo Barcelona (Unknown); Biomechanical Engineering Lab (BIOMEC) - Universitat Politècnica de Catalunya (UPC) (Unknown); Institut Nacional d'Educació Física de Catalunya (INEFC) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ABLEexovsKAFO
Record Dates: First submitted 2021-03-25; First posted 2021-04-22 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injury; Exoskeleton; KAFO; Gait; Rehabilitation; Lower-limb; Gait Kinematics; Robotics; Energy Efficiency; Oxygen Consumption; Gas exchange; Neurorehabilitation; Paraplegia; Walking; Passive orthoses; Assistive technology; Usability; Randomized crossover
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia

STUDY DESIGN:
Intervention Model Description: Participants will complete 10 gait training sessions during a 5-week period with one of the two devices (ABLE Exoskeleton or KAFO orthoses) followed by a post-training assessment. After the training program with the first device, participants will have 2 weeks resting time, after which they will repeat the process with the other device. The initial device assignment (ABLE Exoskeleton or KAFO) is performed randomly.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABLE Exoskeleton - KAFO (Experimental): Participants belonging to this arm start the study by performing the training program using the ABLE Exoskeleton. After the resting period, they repeat the training program using KAFO orthoses.
  Interventions: Device: ABLE Exoskeleton; Device: KAFO Orthosis
- KAFO - ABLE Exoskeleton (Experimental): Participants belonging to this arm start the study by performing the training program using the KAFO orthoses. After the resting period, they repeat the training program using the ABLE Exoskeleton.
  Interventions: Device: ABLE Exoskeleton; Device: KAFO Orthosis

INTERVENTIONS:
Device: ABLE Exoskeleton — Participants will use the ABLE Exoskeleton to perform therapy activities (sit-to-stand transfers, walk, turns, balance exercises, normalized tests). Participants will perform a total of 10 training sessions of an approximate duration of 90 minutes.
Device: KAFO Orthosis — Participants will use a pair of KAFO-type passive orthosis to perform therapy activities (sit-to-stand transfers, walk, turns, balance exercises, normalized tests). Participants will perform a total of 10 training sessions of an approximate duration of 90 minutes.

SUMMARY:
This randomized crossover study will compare walking with KAFO type orthoses (current standard of care) versus the ABLE Exoskeleton device, during walking in patients with spinal cord injury in a hospital setting. The ABLE Exoskeleton is a robotic exoskeleton that actively assists individuals with mobility problems to stand up, walk and sit down.

The main objective of the study is to compare the energy efficiency during gait with both devices. Secondary objectives are: compare gait kinematics, usability, user's satisfaction, physical activity and psychosocial impact. The study will also serve to evaluate the usability and safety of the ABLE Exoskeleton in clinical practice.

Subjects will complete 10 gait training sessions during a 5-week period with 1 of the 2 devices randomly selected, followed by a post-training assessment consisting of 1 session. Once the test is completed, subjects will have a 2-week rest period after which they will repeat the process with the other device for 5 weeks (followed by 1 post-training assessment session). The study will be conducted at Hospital Asepeyo Barcelona in Spain, where a total of 10 patients will be recruited.

DETAILED DESCRIPTION:
The primary objective of this study is determining the energy efficiency through gases exchange and kinematic gait analysis to compare the standard of assistance (KAFO type orthoses) and the ABLE Exoskeleton, a robotic gait assistance device, in patients with spinal cord injury (SCI) in a hospital setting.

The secondary objectives are to compare the performance of KAFO-type orthoses with that of the ABLE Exoskeleton device by:

* Kinematic analysis of gait and spatiotemporal gait parameters.
* Evaluation of the time and effort required to learn to use the device (usability).
* Evaluation of the impact that physical activity has on participants after gait training.
* Evaluation of the level of satisfaction of the participants.

In addition to these objectives, the safety of the ABLE Exoskeleton as an assistive device for gait rehabilitation in SCI patients will be evaluated throughout the study.

Participants will perform 2 training sessions per week of approximately 90 minutes duration for 5 weeks with each of the devices, completing a total of 10 sessions with KAFO type orthoses and 10 sessions with the ABLE Exoskeleton. Before starting the training period, the physical capacity of the participants will be measured. During the training period sessions, different measurements of the level of assistance, spatiotemporal gait variables and usability will be taken. Standardized clinical assessments will also be performed during sessions 5 and 10 (assessment sessions). At the end of the training period, a post-training assessment will be performed, consisting of 1 session where the physical capacity of the participants will be measured. After finishing the training period with one of the devices, participants will have a rest period of 2 weeks, after which they will change devices and repeat the whole process.

The main hypothesis of the study is that gait efficiency in patients with SCI is improved (lower energy consumption) when using the ABLE Exoskeleton device in comparison with KAFO-type orthoses. The increase in gait efficiency encourages patients to stand and walk for longer periods instead of using the wheelchair, which boosts their rehabilitation and improves their health.

Secondary hypotheses are:

* The ABLE Exoskeleton device will improve the kinematics and spatiotemporal parameters of gait (more closely resemble the gait pattern of a healthy individual), relative to KAFO-type orthoses.
* The ABLE Exoskeleton device will have a more positive impact on the mobility and psychosocial health of participants with SCI in the study, with respect to KAFO-type orthoses.
* The ABLE Exoskeleton device is a safe device to use in a hospital setting as an assistive device during gait rehabilitation in SCI patients.

ELIGIBILITY:
Inclusion Criteria:

* From 18 to 70 years old
* Chronic or subacute spinal cord injury.
* Currently in treatment as in-patient or ambulatory in the investigational site.
* From AIS A to AIS D with enough arm strength to withstand the bodyweight in a walking frame.
* Previous experience walking with KAFO orthoses (must tolerate standing).
* Ability to give informed consent

Exclusion Criteria:

* WISCI II >16 without the exoskeleton.
* 5 or more fragility fracture risk factors according to Craven et al.
* History of fragility fractures of lower limbs in the past 2 years.
* Deterioration > 3 points of the total International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) motor score within the last 4 weeks.
* Spinal instability
* Modified Ashworth scale (MAS) > 3 in lower limbs
* Unable to tolerate 30 minutes standing without clinical symptoms of orthostatic hypotension.
* Unable to walk 5 meters with KAFO orthoses and the support of a walking frame with wheels.
* Psychological or cognitive issues that do not allow a participant to follow the study procedures.
* Any neurological condition other than SCI
* Medically unstable
* Severe comorbidities including any condition that a physician considers to not be appropriate to complete participation in the study.
* Ongoing skin issues
* Height, width, weight or other anatomical constraints (such as leg length differences) incompatible with the device
* Insufficient Range of Motion (ROM) for ABLE Exoskeleton device
* Known pregnancy or breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-09-17 (Actual)

PRIMARY OUTCOMES:
Measurement of gas exchange during 6 Minute Walk Test (6 MWT) | Session #5, Session #10. Sessions take place 2x/week over a 5 week training period.
  6 Minute Walk Test (6 MWT) measures the distance a person can walk in 6 minutes. There are different possibilities for performing this test. For this study, we will use a track of at least 10 meters, where patients walk back and forth.
Measurement of gas exchange during the Timed Up and Go Test (TUG) | Session #5, Session #10. Sessions take place 2x/week over a 5 week training period.
  Timed Up and Go Test (TUG) measures the time it takes a person to get up from a chair, walk 3 meters, turn around and sit down again. It is a widely used test to assess balance and the risk of falls in different patient groups.
Measurement of gas exchange during Graded exercise testing (GXT) | Change from preliminary assessment through study completion, an average of 16 weeks.
  Maximal Graded Exercise Test (GXT) is a screening tool to track an individual's fitness level. The test evaluates the participant's exercise capacity by measuring the cardiovascular response to physical activity. Through this test, the values of maximal oxygen consumption will be obtained and used to obtain metrics to assess energy efficiency during the gait.
Measurement of gas exchange during 10 Meter Walk Test (10MWT) | Session #5, Session #10. Sessions take place 2x/week over a 5 week training period.
  The 10 Meter Walk Test (10 MWT) measures the time a person needs to walk 10 meters. The test is performed with a dynamic (flying) start with two-meter acceleration, a timed ten-meter distance and two-meter deceleration.

SECONDARY OUTCOMES:
Measurement of the Level of Assistance to perform therapy activities. | Up to 5 weeks
  To measure the time required to learn to use the device under investigation, different activities (don/doff, balance, walking, advanced abilities) will be performed during the training period. The difficulty of each activity increases as they are completed.
Perceived level of exertion | Up to 6 weeks
  For measuring impact on the perceived level of exertion, the BORG will be tested after the 6 MWT/TUG/GXT with and without the device. The BORG scale measures the subjective level of intensity in physical work on a 15-grade scale. It ranges from 6 (No exertion at all) to 20 (Maximal exertion).
Fatigue Visual Analog Scale (VAS) | Up to 6 weeks
  The scale consists of a straight line where one end means the absence of fatigue and the other end means maximal fatigue. The patient selects a point in the line which coincides with their level of fatigue.
Spinal Cord Independence Measure (SCIM) III | Up to 10 days before first session and up to 10 days after first session
  Spinal Cord Independence Measure (SCIM III) scale focuses on the ability to perform activities of daily living in persons with SCI. The SCIM III consists of three subscales: Self-Care, Respiratory and Sphincter Management, Mobility (room and toilet) and Mobility (indoors and outdoors, on even surface). A total score of 0 (totally dependent) to 100 (totally independent) points can be achieved.
Quebec User Evaluation of Satisfaction with assistive Technology (QUEST 2.0) | Up to 6 weeks
  QUEST 2.0 is designed to measure the level of satisfaction and the value people attribute to assistive technologies. It does so using 12 variables which are scored on a 5 point scale in terms of perceived importance and satisfaction. While items 1-8 rate the satisfaction with the device, items 9-12 are for assessing the satisfaction with the service. If the users are not very satisfied with a feature, they are asked to provide specific feedback. The final score is the mean sum scores of all valid responses with a range of 1 (not satisfied at all) to 5 (very satisfied).
Psychosocial Impact of Assistive Devices Scales (PIADS) | Up to 6 weeks and followup (4 weeks after study completion).
  PIADS is a 26-item (7-point Likert-Scale), self-report questionnaire designed to assess the effects of an assistive device on functional independence, well-being, and quality of life. It is divided into three subscales: Competence, adaptability and self-esteem. For each of the subscales, typically means are calculated that range from -3 (maximum negative impact) to +3 (maximum positive impact). To have only positive sum scores, the range of the individual scores are shifted to 1 to 7, meaning that the sum scores range from 1 *26 (26, maximum negative impact) to 7 *26 (182, maximum positive impact). The PIADS is a responsive measure and sensitive to important variables such as the user's clinical condition, device stigma, and functional features of the device. It has been shown to accurately reflect the self-described experiences of people who use assistive devices.

OTHER OUTCOMES:
Gait Analysis | Session #5, Session #10. Sessions take place 2x/week over a 5 week training period.
  Kinematic and kinetic gait parameters will be calculated from data acquired with a motion capture system.

CONTACTS AND LOCATIONS:
Overall Officials: Lluís Guirao Cano, MD PhD, Principal Investigator — Hospital ASEPEYO Sant Cugat
Locations (1):
- Hospital Asepeyo Sant Cugat, Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No